CLINICAL TRIAL: NCT03337854
Title: Analysis With Clusters of QUAntitative Tomodensitometric Vascular, bronchIal and Parenchymal Pulmonary Parameters for COPD Patients
Acronym: ACQUAVIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Transitionnal Research International Laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017/44
Record Dates: First submitted 2017-10-24; First posted 2017-11-09 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: prognostic; phenotype; Computed tomography; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is caused by tobacco consumption. The goal is to characterize on clinical and radiological data, using computed tomography, this illness in order to improve diagnostic and be able to evaluate the prognostic of each patient.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by emphysematous destruction of pulmonary parenchyma, airway obstruction that participate in chronic temporary obstruction of airways. COPD has multiple clinical presentations that define phenotypes but doesn't take into account those anatomo-pathologic modifications. Moreover, the prognostic interest of those structural alteration is unknown. Until now, only PFT allowed to define the severity of the disease, whereas multiple others tools may be useful, such as, symptoms scores, exacerbation frequencies, denutrition. Those structural alterations are available using computed tomography (CT), that may also have an interest in prognostic or in treatment follow- up.

CT is widely used in clinical practice for COPD patients at basal state and in exacerbations. Quantitative CT is able to combine acquisition of objective and reproductible informations on parenchymal destruction (emphysema), bronchial wall remodeling, and pulmonary vessels alteration. The investigators' team developed software tools to determine quantitative structural modifications of airways, emphysema and small pulmonary vessels1,2.

The team has been able to build a score "Paw score" combining PaO2 with CT parameters of bronchial wall thickness and small pulmonary vessels percentage2. This score allowed to predict the presence of severe pulmonary hypertension in patients with COPD. Pulmonary hypertension is a complication of COPD that increase morbi-mortality.

The hypothesis is that morphological quantitative analysis combined with structural alterations of airways has a prognostic interest.

The main goal is to determine morphological phenotypes of COPD using a cluster analysis combining emphysema, bronchial wall thickness and pulmonary vessels.

The other main goal is to predict evolution of COPD patients based on clinical outcomes (exacerbations frequency, mortality, mMRC, SGQLQ) and lung function testing (decline in FEV-1 TLCO, PaO2).

The team also wants to analyze clinical data of survival, exacerbation and symptoms in following years of the CT of each cluster in historic-prospective way.

The secondary goals are to describe clinical, functional and biological clusters. Analyse of correlations will be studied. Moreover, we will investigate the interest of the "Paw score" as a prognostic marker and as a correlated parameter.

This is a retrospective study. We want to take information from the year before CT, to the year after CT. At the date of the consultation concomitant with CT we want to know all the clinical, functional and biological data of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Inhalated toxic exposure:

  * Tobacco exposure (present or past, over 10 pack years)
  * And/or professional exposure to a toxic
* Obstructive syndrome with a FEV1/FVC ≤ 0.7 after inhalation of a bronchodilatator and measured at stable state (without exacerbation)
* Computed tomography performed without injection contrast during common care

Exclusion Criteria:

* Patients with an exacerbation within 6 weeks before computed tomography
* Artefacts movements on computed tomography incompatible with quantitative analyse
* Broncho-pulmonary cancer (old or present)
* History of pulmonary surgery
* No follow-up for 1 year after scan
* Opposition of the patient to the use of his data (clinical, functional and imaging).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with an age ≥ 40 years and inhalated toxic exposure like Tobacco exposure (present or past, over 10 pack years) and/or professional exposure to a toxic, in presence of obstructive syndrome with a FEV1/FVC ≤ 0.7 after inhalation of a bronchodilatator and measured at stable state (without exacerbation).
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Phenotypes of Chronic obstructive pulmonary disease (COPD) | Day 1
  Measure of emphysema
Phenotypes of Chronic obstructive pulmonary disease (COPD) | Day 1
  Measure of proximal bronchial wall thickness
Phenotypes of Chronic obstructive pulmonary disease (COPD) | Day 1
  Measure of dimensions of the pulmonary arteries
Phenotypes of Chronic obstructive pulmonary disease (COPD) | Day 1
  Measure of ratio of main pulmonary artery over aoarta diameter

SECONDARY OUTCOMES:
Clinical data of survival | Day 1
  Date of death
Exacerbations | Day 1
  Number of exacerbations

OTHER OUTCOMES:
Number of pack per year of tobacco | Day 1
  Number of pack per year of tobacco
Clinical scores | Day 1
  Score COPDAssessmentTest "CAT" Scale range: minimum value: 0, maximum value: 40. Only total score is reported. Higher values are considered to be bad outcome. Subscale are not reported, but there are combined by summed to compute the total score.
Clinical scores | Day 1
  Score St Georges Scale range: minimum value: 0, maximum value: 3989.4. Only total score is reported. Higher values are considered to be bad outcome. Subscale (symptoms, activities, impact) are not reported, but there are combined by summed to compute the total score.
Clinical scores | Day 1
  Score mMRC (Medical Research Council ) Scale range: minimum value: 0, maximum value: 4. Only total score is reported. Higher values are considered to be bad outcome.
Clinical scores | Day 1
  Score Global Initiative for Chronic Obstructive Lung Disease (GOLD) Scale range: minimum value: 0, maximum value: 4. Only total score is reported. Higher values are considered to be bad outcome.
Clinical data | Day 1
  Six minute walk test (meters, and % predicted)
Pulmonary function test | Day 1
  Forced Expiratory Volume - FEV1 (L)
Pulmonary function test | Day 1
  Forced Expiratory Volume/ Forced Volume Capacity (FEV1/FVC)(%)
Pulmonary function test | Day 1
  value of KCO (Carbon Monoxide Diffusing Capacity (DLCO) divided by Alveolar Volume(VA))
Pulmonary function test | Day 1
  transfer factor of the lung for carbon monoxide (TLCO)
Pulmonary function test | Day 1
  total lung capacity (TLC)
Arterial blood gazes | Day1
  pH
Arterial blood gazes | Day1
  Partial pressure of oxygen in arterial blood (PaO2) in mmHg
Arterial blood gazes | Day1
  Partial pressure of carbon dioxide in arterial blood in mmHg.
Arterial blood gazes | Day1
  Hemoglobin (g/dL)
Arterial blood gazes | Day1
  carboxyhemoglobin (%)
Biology | Day1
  C-reactive protein; cross-reacting protein (mg/l).
Biology | Day1
  α1-antitrypsin (mg/l).
Clinical parameter | Day1
  weight (kilograms)
Clinical parameter | Day1
  Height (meters)
Clinical parameter | Day1
  comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: François LAURENT, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France